CLINICAL TRIAL: NCT05432050
Title: Bispectral Index and Patient State Index During General Anesthesia With Remimazolam: a Prospective Observational Study
Brief Title: Bispectral Index and Patient State Index During General Anesthesia With Remimazolam
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: H-2204-008-1313
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Remimazolam; Anesthesia, General; Hypnotics and Sedatives; Thyroid Disease; Breast Diseases; Parathyroid Diseases
Keywords: Patient state index; Bispectral index; Electroencephalography
MeSH Terms: conditions — Thyroid Diseases; Breast Diseases; Parathyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remimazolam anesthesia: General anesthesia will be induced and maintained by remimazolam and the depth of anesthesia will be monitored with both the bispectral index and patient state index at the same time.
  Interventions: Device: Bispectral index and Patient state index monitoring

INTERVENTIONS:
Device: Bispectral index and Patient state index monitoring — The depth of anesthesia will be monitored with both the bispectral index and patient state index at the same time.

SUMMARY:
The aim of this study is to compare the bispectral index (BIS) and patient state index (PSI) during general anesthesia using remimazolam. The infusion rate of remimazolam is 6-12mg/kg/h during induction of anesthesia and 1-2mg/kg/h during maintenance of anesthesia. To calculate the fraction, the sum of times when BIS<60 and PSI <50 will be divided by the time from the loss of consciousness during induction of anesthesia to fully awake during emergence. We will compare the fraction of BIS <60 and the fraction of PSI <50 to find if there is some difference between the two depth of anesthesia monitoring devices during remimazolam anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years need general anesthesia
* American Society of Anesthesiologists (ASA) Classification I, II
* Written informed consent

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Classification III, IV, V
* BMI > 40kg/m^2
* Past medical history of anaphylactic reaction to remimazolam, remifentanil, or other benzodiazepines.
* Administration of anxiolytics, antipsychotics, rifampicin, succinylcholine, neostigmine, flumazenil, and cyclosporin within the past 24 hours
* Benzodiazepine user (e.g. for seizure control)
* Transfer to intensive care unit after surgery

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (ASA class I,II) who need general anesthesia for surger
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of time when bispectral index (BIS) was < 60 | During anesthesia (up to 6hours)
  The percentage of time when BIS was < 60 (divided by the time between the loss of consciousness during induction of anesthesia and the full awakening during emergence from anesthesia.)
The percentage of time when patient state index (PSI) was < 50 | During anesthesia (up to 6hours)
  The percentage of time when PSI was < 50 (divided by the time between the loss of consciousness during induction of anesthesia and the full awakening during emergence from anesthesia.)

SECONDARY OUTCOMES:
Heart rate (bpm) | During anesthesia (up to 6hours)
  Heart rate (bpm) measured before induction of anesthesia, at loss of consciousness, and before transfer to post-anesthesia care unit.
blood pressure (mmHg) | During anesthesia (up to 6hours)
  blood pressure (mmHg) measured before induction of anesthesia, at loss of consciousness, and before transfer to post-anesthesia care unit.
Bispectral index (BIS) during anesthesia | During anesthesia (up to 6hours)
  Bispectral index (BIS) is continuously recorded during anesthesia.
Patient state index (PSI) during anesthesia | During anesthesia (up to 6hours)
  Patient state index (PSI) is continuously recorded during anesthesia.
The percentage of time when bispectral index (BIS) was < 60, and > 40. | During anesthesia (up to 6hours)
  The percentage of time when BIS was < 60, and > 40 (divided by the time between the loss of consciousness during induction of anesthesia and the full awakening during emergence from anesthesia.)
The percentage of time when patient state index (PSI) was < 50, and > 25. | During anesthesia (up to 6hours)
  The percentage of time when PSI was < 50, and > 25 (divided by the time between the loss of consciousness during induction of anesthesia and the full awakening during emergence from anesthesia.)
The last number patient remember that he/she spoke during induction of anesthesia | During anesthesia (up to 6hours)
  The last number patient remember that he/she spoke during induction of anesthesia (begin from 1 to loss of consciousness)
Remimazolam infusion history | During anesthesia (up to 6hours)
  The rate of Remimazolam infusion is recorded during anesthesia.
Remifentanil infusion history | During anesthesia (up to 6hours)
  The target effect-site concentration of remifentanil infusion is recorded during anesthesia.
Total amount of remimazolam used (mg/kg/h) | During anesthesia (up to 6hours)
  Total amount of remimazolam used (mg/kg/h) during anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD,PhD, Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sneyd JR, Gambus PL, Rigby-Jones AE. Current status of perioperative hypnotics, role of benzodiazepines, and the case for remimazolam: a narrative review. Br J Anaesth. 2021 Jul;127(1):41-55. doi: 10.1016/j.bja.2021.03.028. Epub 2021 May 6. PMID 33965206
- [Background] Masui K. Remimazolam besilate, a benzodiazepine, has been approved for general anesthesia!! J Anesth. 2020 Aug;34(4):479-482. doi: 10.1007/s00540-020-02755-1. Epub 2020 Mar 10. No abstract available. PMID 32157465
- [Background] Sneyd JR, Rigby-Jones AE. Remimazolam for anaesthesia or sedation. Curr Opin Anaesthesiol. 2020 Aug;33(4):506-511. doi: 10.1097/ACO.0000000000000877. PMID 32530890
- [Background] Schuttler J, Eisenried A, Lerch M, Fechner J, Jeleazcov C, Ihmsen H. Pharmacokinetics and Pharmacodynamics of Remimazolam (CNS 7056) after Continuous Infusion in Healthy Male Volunteers: Part I. Pharmacokinetics and Clinical Pharmacodynamics. Anesthesiology. 2020 Apr;132(4):636-651. doi: 10.1097/ALN.0000000000003103. PMID 31972655
- [Background] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555